CLINICAL TRIAL: NCT00079833
Title: A Phase III, Multicenter, Open-Label Study To Evaluate the Control of Gastric Acid Secretion With Esomeprazole In Patients With Gastric Acid Hypersecretory States Including Idiopathic Hypersecretion and Zollinger-Ellison Syndrome For 12 Months
Brief Title: Esomeprazole In Patients With Gastric Acid Hypersecretory States Including Idiopathic Hypersecretion and Zollinger-Ellison Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D9612C00025
Record Dates: First submitted 2004-03-16; First posted 2004-03-17 (Estimated); Last update posted 2010-11-19 (Estimated); Status verified 2010-11

CONDITIONS: Zollinger-Ellison Syndrome
Keywords: gastric acid hypersecretory conditions; Idiopathic Hypersecretion; Excessive Gastric Acid secretion
MeSH Terms: conditions — Zollinger-Ellison Syndrome | interventions — Esomeprazole

INTERVENTIONS:
Drug: Esomeprazole magnesium (Nexium)

SUMMARY:
This research study will determine if esomeprazole, when administered twice daily at 40, 80, or 120 mg doses, can control excessive stomach acid secretion.

ELIGIBILITY:
Inclusion Criteria:

* Males or females at least 18 years of age.
* Diagnosis of Zollinger-Ellison Syndrome or idiopathic hypersecretion

Exclusion Criteria:

* Pregnant or lactating females
* History of drug addiction or alcohol abuse within 12 months prior to Screening.
* History of intolerance to any proton pump inhibitors or any ingredient in their formulation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25
Dates: Start 2003-11; Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
To assess the gastric acid secretory rate at the final study visit.
Control is defined as gastric acid secretory rate below 10 mEq/h or below 5 meq/h for patients with prior gastric acid reducing Surgery

SECONDARY OUTCOMES:
The status (controlled or not controlled) of gastric acid secretory rate at the Month 6 study visit.
Control is defined as gastric acid secretory rate below 10 mEq/h or below 5 meq/h for patients with prior gastric acid reducing surgery.
The following safety variables will be assessed at Month 6 and Month 12: adverse events, clinical laboratory results (ie, chemistry, hematology, urinalysis), physical examinations, and EGDs.

CONTACTS AND LOCATIONS:
Overall Officials: Nexium Medical Science Director, MD, Study Director — AstraZeneca
Locations (8):
- United States (5):
  - Research Site, Los Angeles, California
  - Research Site, Gainesville, Florida
  - Research Site, Columbus, Ohio
  - Research Site, King of Prussia, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
- France (3):
  - Research Site, Clichy
  - Research Site, Paris
  - Research Site, Saint-Germain-en-Laye